CLINICAL TRIAL: NCT04324736
Title: "Coronavirus SARS-CoV2 and Diabetes Outcomes" : CORONADO
Brief Title: "COVID-19 and Diabetes Outcomes"
Acronym: CORONADO
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC20_0148
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Coronavirus; Diabetes
MeSH Terms: conditions — Coronavirus Infections; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with diabetes
  Interventions: Other: no interventional study
- Patients without diabetes
  Interventions: Other: no interventional study

INTERVENTIONS:
Other: no interventional study — no interventional study

SUMMARY:
COVID-19 (Coronavirus Disease-2019) is a life-threatening infectious disease caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) that appeared in December 2019 in the Wuhan district. COVID-19 has since affected more than 150 countries across the world and especially France. The first epidemiological data, mostly from Chinese studies, indicate that diabetes is one of the most common comorbidities, with high blood pressure, in patients with COVID-19. Moreover, the presence of diabetes at admission would be a risk factor for both ICU hospitalization and death.

Nevertheless, specific data on people with diabetes and COVID-19 are fragmentary, justifying the achievement of a dedicated prospective observational study.

The French nationwide CORONADO study aims to specifically describe the phenotypic characteristics of patients with diabetes admitted to hospital with COVID-19 infection. Particular attention will be devoted to glycemic control at admission (i.e. the level of HbA1c), the diabetic complications, as well as anti-diabetic and antihypertensive therapies.

This study will provide answers to caregivers and patients with diabetes regarding the risk factors related to diabetes for COVID-19 prognosis. This pilot study will be used for the development of new studies and for the establishment of recommendations for the cost of care in patients with diabetes and COVID-19.

ELIGIBILITY:
Inclusion criteria

* Patients admitted in a hospital center since 10th march 2020
* Patients with COVID19 with biological proof (specific PCR) or with clinical and radiological diagnosis.
* Patient with diabetes known before the admission
* New onset diabetes discovered at admission (HbA1c value strictly greater than 6.5%)

exclusion criteria

* subjects opposed to the use of their data
* minors, adults under guardianship, protected persons
* subject having already been included in the CORONADO study (subject readmitted after discharge following the initial stay). Only the data of the first stay will be maintained.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: diabetic patients treated for COVID-19 in a hospital center and non diabetic patients treated for COVID-19 in a hospital center
Sampling Method: Probability Sample
Enrollment: 5309 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Assess the prevalence of severe forms among hospitalized patients with diabètes and COVID-19 | 1 month
  Prevalence of severe forms among all COVID-19 patients with diabetes

SECONDARY OUTCOMES:
describe the clinical and biological characteristics of hospitalized subjects with diabetes and COVID-19 | 1 month
  Use the body weight, type of diabetes, tglycemic control (HbA1C at admission), the comorbidities and complications associated with diabetes and finally the usual therapies.
describe the prognosis of hospitalized subjects with diabetes and COVID-19 | 1 month
  death at 7 days after admission, hospital death and date of death, total length of hospitalization and discharge procedures, serious form requiring the use of artificial ventilation with tracheal intubation and date of use of this treatment, decision to limit
describe the care management of hospitalized subjects with diabetes and COVID-19 | 1 month
  care service where the patient is taken care of, insulin therapy (IVSE or multi-injection) and dose of insulin required on D2 and D7

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cariou B, Wargny M, Boureau AS, Smati S, Tramunt B, Desailloud R, Lebeault M, Amadou C, Ancelle D, Balkau B, Bordier L, Borot S, Bourgeon M, Bourron O, Cosson E, Eisinger M, Gonfroy-Leymarie C, Julla JB, Marchand L, Meyer L, Seret-Begue D, Simon D, Sultan A, Thivolet C, Vambergue A, Vatier C, Winiszewski P, Saulnier PJ, Bauduceau B, Gourdy P, Hadjadj S; CORONADO investigators. Impact of diabetes on COVID-19 prognosis beyond comorbidity burden: the CORONADO initiative. Diabetologia. 2022 Sep;65(9):1436-1449. doi: 10.1007/s00125-022-05734-1. Epub 2022 Jun 15. PMID 35701673
- [Derived] Tramunt B, Smati S, Coudol S, Wargny M, Pichelin M, Guyomarch B, Al-Salameh A, Amadou C, Barraud S, Bigot E, Bordier L, Borot S, Bourgeon M, Bourron O, Charriere S, Chevalier N, Cosson E, Feve B, Flaus-Furmaniuk A, Fontaine P, Galioot A, Gonfroy-Leymarie C, Guerci B, Lablanche S, Lalau JD, Larger E, Lasbleiz A, Laviolle B, Marre M, Munch M, Potier L, Prevost G, Renard E, Reznik Y, Seret-Begue D, Sibilia P, Thuillier P, Verges B, Gautier JF, Hadjadj S, Cariou B, Mauvais-Jarvis F, Gourdy P. Sex disparities in COVID-19 outcomes of inpatients with diabetes: insights from the CORONADO study. Eur J Endocrinol. 2021 Jul 5;185(2):299-311. doi: 10.1530/EJE-21-0068. PMID 34085949
- [Derived] Wargny M, Potier L, Gourdy P, Pichelin M, Amadou C, Benhamou PY, Bonnet JB, Bordier L, Bourron O, Chaumeil C, Chevalier N, Darmon P, Delenne B, Demarsy D, Dumas M, Dupuy O, Flaus-Furmaniuk A, Gautier JF, Guedj AM, Jeandidier N, Larger E, Le Berre JP, Lungo M, Montanier N, Moulin P, Plat F, Rigalleau V, Robert R, Seret-Begue D, Serusclat P, Smati S, Thebaut JF, Tramunt B, Vatier C, Velayoudom FL, Verges B, Winiszewski P, Zabulon A, Gourraud PA, Roussel R, Cariou B, Hadjadj S; CORONADO investigators. Predictors of hospital discharge and mortality in patients with diabetes and COVID-19: updated results from the nationwide CORONADO study. Diabetologia. 2021 Apr;64(4):778-794. doi: 10.1007/s00125-020-05351-w. Epub 2021 Feb 17. PMID 33599800
- [Derived] Wargny M, Gourdy P, Ludwig L, Seret-Begue D, Bourron O, Darmon P, Amadou C, Pichelin M, Potier L, Thivolet C, Gautier JF, Hadjadj S, Cariou B; CORONADO investigators. Type 1 Diabetes in People Hospitalized for COVID-19: New Insights From the CORONADO Study. Diabetes Care. 2020 Nov;43(11):e174-e177. doi: 10.2337/dc20-1217. Epub 2020 Aug 26. No abstract available. PMID 32847826
- [Derived] Cariou B, Hadjadj S, Wargny M, Pichelin M, Al-Salameh A, Allix I, Amadou C, Arnault G, Baudoux F, Bauduceau B, Borot S, Bourgeon-Ghittori M, Bourron O, Boutoille D, Cazenave-Roblot F, Chaumeil C, Cosson E, Coudol S, Darmon P, Disse E, Ducet-Boiffard A, Gaborit B, Joubert M, Kerlan V, Laviolle B, Marchand L, Meyer L, Potier L, Prevost G, Riveline JP, Robert R, Saulnier PJ, Sultan A, Thebaut JF, Thivolet C, Tramunt B, Vatier C, Roussel R, Gautier JF, Gourdy P; CORONADO investigators. Phenotypic characteristics and prognosis of inpatients with COVID-19 and diabetes: the CORONADO study. Diabetologia. 2020 Aug;63(8):1500-1515. doi: 10.1007/s00125-020-05180-x. Epub 2020 May 29. PMID 32472191